CLINICAL TRIAL: NCT06017765
Title: Coping After Loss Through Mindfulness Training in Grieving Adults With Prolonged Grief Disorder - A Neuroimaging Pilot Study
Brief Title: Coping After Loss Through Mindfulness in Adults With Prolonged Grief Disorder
Acronym: CALM-NiPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: Northeastern University (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Cyceron (Unknown); Université de Caen Normandie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 22-0245; 2022-A02603-40 (Registry Identifier: ANSM ID-RCB)
Record Dates: First submitted 2023-07-20; First posted 2023-08-30 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Prolonged Grief Disorder
Keywords: Prolonged Grief Disorder; Bereavement; Mindfulness Training; Script-driven Imagery; Stress Reactivity; Neuroimaging
MeSH Terms: conditions — Prolonged Grief Disorder | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: The study model is a pilot randomized waitlist controlled trial of an 8-session mindfulness training program (i.e., Stress Management and Resiliency Training, SMART program) delivered weekly for Prolonged Grief Disorder, either within 4 weeks (immediate) or after 12 weeks (waitlist). After participants have completed the baseline assessment (V0), they will be randomly assigned (1:1 randomization) to either the immediate mindfulness training group or the waitlist control group. The waitlist control group will wait for 12 weeks (when the immediate intervention group finished all study procedures, including the follow-up assessment) before receiving the mindfulness training, which is the same intervention as employed in the immediate intervention group.
Who Masked: Outcomes Assessor
Masking Description: Participants will be assessed for psychiatric symptoms (primary objective) by blinded Independent Evaluators, who will not be involved in the mindfulness training sessions. Participants will be instructed to keep their evaluators blinded to the randomization. Blinded Independent Evaluators will be clinical psychologists who are fully trained in assessing the different measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Meditation Training group (Experimental): The Immediate Meditation Training group will immediately receive 8 weekly sessions of Mindfulness Training within 4 weeks after the Baseline visit (V0, during which participants are randomized).
  Interventions: Behavioral: Meditation Training
- Waitlist Control group (Other): The Waitlist Control group will receive the Mindfulness Training after a waiting time of 12 weeks. Participants in this group will not receive any type of intervention before this and will wait till the Immediate Meditation Training group finished all assessment visits (including the follow-up visit in week 12 (V3)).
  Interventions: Behavioral: Waitlist

INTERVENTIONS:
Behavioral: Meditation Training — The Meditation Training consists of 8 weekly sessions of Mindfulness Training and is adapted from the group-based Stress Management and Resiliency Training - Relaxation Response Resiliency Program, SMART-3RP. This training is structured around the following four goals:
  1. Education about stress response
  2. Elicitation of the Relaxation Response through Mindfulness Training
  3. Creating adaptive perspectives
  4. Coping strategiest.
  Other Names: Mindfulness Training; SMART
  Arms: Immediate Meditation Training group
Behavioral: Waitlist — The waitlist consists of a waiting time of 12 weeks during which participants will nog receive any type of intervention.
  Arms: Waitlist Control group

SUMMARY:
The goal of this clinical trial is to pilot the effectiveness of an 8-week standardized Mindfulness Training program to decrease the psychiatric and somatic symptoms of prolonged grief disorder (PGD) and to examine changes in physiological and neuroimaging biomarkers of bereavement-related stress reactivity that are associated with Mindfulness Training in grieving adult patients (men and women, aged 18-60) who are diagnosed with PGD.

The main questions it aims to answer are:

1. What is the effectiveness of Mindfulness Training to lower PGD symptom severity?
2. What is the effectiveness of Mindfulness Training on physiological and neuroimaging biomarkers of stress reactivity?
3. What are the potential mechanisms of treatment change of Mindfulness Training?

Participants will be:

* randomly assigned to immediately receiving an 8-week Mindfulness Training program or after a 12-week waitlist.
* assessed for psychiatric and somatic symptoms and for physiological responses during a baseline, midpoint and endpoint visit, and at a one-month follow-up visit.
* assessed for functional neuroimaging biomarkers of bereavement-related and general stress reactivity at the baseline and endpoint visits using a script-driven imagery task (which induces bereavement-related stress reactivity during an imagery of a personal situation related to the death compared to imagery of a neutral personal situation), and loud tones stress task (which induces general stress reactivity).

Researchers will compare the Mindfulness Training group (which consists of patients with PGD who will receive the Mindfulness Training immediately) with the waitlist control group (which consists of patients with PGD who are waiting on a waitlist to receive the training after the Mindfulness Training group) to investigate if they differ in PGD symptom severity as well as physiological and neuroimaging biomarkers of stress reactivity.

DETAILED DESCRIPTION:
Bereavement is a major life stressor that triggers a stress response that can last months or years after the death of a loved one. This condition of persisting grief response called Prolonged Grief Disorder (PGD) has been recently included in the World Health Organization (WHO) International Classification of Diseases, and the fifth text-revised version of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5TR). A core symptom of PGD is the heightened reactivity to reminders of the death. This stress response, if exaggerated and persisting, is associated with increased risk for mental health problems including suicide, as well as somatic problems such as cardiac adverse events. To date, no efficacious intervention for reducing a bereavement-related stress response exist to prevent the negative health outcomes of adults who lost a loved one. Mindfulness Training has shown efficacy to decrease the general stress reactivity, as was shown in healthy individuals and in anxiety disorders, supposedly by improving emotional regulation. Therefore, it has the potential to successfully target bereavement-related stress-reactivity in grievers, as supported by our pilot data. However, it is unknown whether mindfulness meditation may also decrease bereavement-specific stress reactivity, one of the core symptoms of PGD. Furthermore, little is known about the neurobiological changes that underlie the decrease in stress reactivity that results from mindfulness training.

The present proposal is the first ever clinical trial to pilot the effectiveness of an 8-week Mindfulness Training to decrease psychiatric and somatic symptoms of PGD in adult patients, as well as to pilot changes in physiological and neuroimaging biomarkers of bereavement-related stress reactivity that are associated with Mindfulness Training using a script-driven imagery task (which induces bereavement-related stress reactivity during an imagery of a personal situation related to the death compared to imagery of a neutral personal situation), and loud tones stress task (which induces general stress reactivity). As PGD is a newly recognized psychiatric condition, there are very limited data available about its pathophysiology and neurobiology, and in particular how treatments can intervene on it. Although mind-body interventions such as Mindfulness Training have recently shown to be effective for stress-related conditions, limited data are available about their mechanisms of actions. Our proposal is the first to examine trauma-related emotional regulation neural circuits implicated in the effects of Mindfulness Training on pathological grief reactions.

1. OBJECTIVES:

   This study aims to examine the effects of an 8-week standardized Mindfulness Training program on PGD symptom severity and stress reactivity, as well as to elucidate the neural mechanism of these effects, in grieving adult patients who are diagnosed with PGD.

   The specific aims of this study are:
   * PRIMARY AIM Aim 1. Examine the efficacy of Mindfulness Training to decrease PGD symptom severity (primary outcome) in a group of patients with PGD who will immediately receive the training versus the waitlist control group consisting of patients with PGD who are waiting on a waitlist to receive the training after the Mindfulness Training group.
   * SECONDARY AIMS Aim 2. Examine the efficacy of Mindfulness Training on physiological and neuroimaging biomarkers of bereavement-related and general stress reactivity in a group of patients with PGD who will immediately receive the training versus the waitlist control group.

   Aim 3. Examine potential mechanisms of action of treatment change of Mindfulness Training in a group of patients with PGD who will immediately receive the training versus the waitlist control group.
2. METHODS:

   The investigators conduct a pilot randomized wait-list controlled trial of an 8-week standardized Mindfulness Training program for PGD and examine its effects on physiological and neural correlates of bereavement-related and general stress reactivity. N=30 adults with PGD are included who will be randomly assigned (1:1 group randomization) to immediately receiving an 8-week Mindfulness Training program (experimental group), adapted from the Stress Management and Resiliency Training - SMART, versus after a 12-week waitlist (control group). During a baseline, midpoint, endpoint, and one-month follow-up visit, participants are assessed for psychiatric and somatic symptoms using several questionnaires. In addition, at the baseline and endpoint visit, the investigators will perform functional magnetic resonance imaging (fMRI) to assess functional neuroimaging biomarkers (brain activity and functional connectivity) of bereavement-related and general stress reactivity while collecting physiological responses (heart rate and skin conductance), using a script-driven imagery task (inducing bereavement-related stress reactivity during imagery of a personal situation related to the death versus imagery of a neutral personal situation), and loud tones stress task (inducing general stress reactivity).

   Participants will not be blinded to the intervention condition. They will complete self-report questionnaires and be assessed by blinded Independent Evaluators, who will not be involved in the Mindfulness Training sessions, at the baseline (week 0), midpoint (week 4), endpoint (week 8), and follow-up visit (week 12). Participants will be instructed to keep their evaluators blinded to the randomization. Blinded Independent Evaluators will be clinical psychologists who are fully trained in the different measures.
3. HYPOTHESES:

   1. Hypothesis 1. It is hypothesized that adult patients with PGD who are assigned to immediate Mindfulness Training will exhibit significantly greater improvements from the baseline to the endpoint visit (and the one-month follow-up visit), than the patients in the waitlist control group, concerning PGD symptom severity (primary outcome), PTSD symptom severity, depressive symptom severity, somatic complaints, and/or the ability to cope with stress, and global symptom improvement and severity.
   2. Hypothesis 2-a. It is hypothesized that adult patients with PGD who are assigned to immediate Mindfulness Training will exhibit significantly greater changes in physiological stress responses, as measured by skin conductance and heart rate,

      * for bereavement-related stress reactivity in response to the imagery of a personal situation related to the death (compared to imagery of a neutral personal situation, using a script-driven imagery task) from the baseline to the endpoint visit, than the patients in the waitlist control group.
      * for general stress reactivity in response (induced by the loud tones stress task) from the baseline to the endpoint visit, than the patients in the waitlist control group.
   3. Hypothesis 2-b. It is hypothesized that adult patients with PGD who are assigned to immediate Mindfulness Training will show significantly greater changes in blood-oxygen-level dependent (BOLD) signals in response to the imagery of a personal situation related to the death (compared to imagery of a neutral personal situation, using a script-driven imagery task) in brain regions that are implicated in emotion regulation and regulatory control at the endpoint visit, compared to the patients in the waitlist control group, including:

      * less BOLD activity in the amygdala,
      * more BOLD activity in the medial prefrontal cortex (consisting of the medial frontal gyrus and rostral anterior cingulate cortex),
      * more functional connectivity between the amygdala and the medial prefrontal cortex.
   4. Hypothesis 3-a. It is hypothesized that at the baseline visit, psychiatric and somatic symptom severity will be significantly correlated with the physiological and neuroimaging biomarkers of bereavement-related stress reactivity in response to the imagery of a personal situation related to the death (compared to imagery of a neutral personal situation).
   5. Hypothesis 3-b. It is hypothesized that greater reductions in psychiatric and somatic symptom severity between the baseline and endpoint visit, will be significantly correlated with greater decreases in physiological and neuroimaging biomarkers of bereavement-specific stress reactivity in response to the imagery of a personal situation related to the death (compared to imagery of a neutral personal situation).
   6. Hypothesis 3-c. It is hypothesized that changes in bereavement-related stress reactivity in response to the imagery of a personal situation related to the death (compared to imagery of a neutral personal situation) will mediate the effects of Mindfulness Training on the reductions in clinical symptom severity.
4. PARTICIPATION:

   - All potential participants are asked to sign the informed consent form (approved by the ethics committee) with a medical doctor/study clinician prior to participation and are given as much time as needed to review the consent form. The consent form states that participation is voluntary, that participants can refuse to answer any questions, that they can withdraw from the research at any time, and that participation in no way impacts their care. All participants must be beneficiaries of the social security system.
5. METHODOLOGY

   1. Power considerations:

      Our primary analysis follows the intention-to-treat (ITT) principle to compare participants' outcomes according to their initial treatment assignment. The investigators restrict the ITT sample to randomized participants who attend at least one treatment session, including those who do not have analyzable neuroimaging and/or psychophysiological data. With N = 30 participants with usable data for aim 2, and alpha = 0.05 (2-tailed), there will be 80% power to detect a large d=1.1 difference.
   2. Dropout and study withdrawal:

   Participants may discontinue their participation if they wish, at any time and for any reason, or upon the decision of the investigator.

   Premature study exits may be (a) progression of the study condition, (b) participants' refusal to continue, (c) withdrawal of consent, (d) protocol violation requiring a study exit, (e) unblinding, (f) by decision of the investigator, (g) by decision of the sponsor, (h) participant non-compliance.

   At every assessment visit, and every 2 weeks during the active phase of the Mindfulness Training, an investigator will assess symptom improvement and worsening, adverse events (reviewed weekly by the Principal Investigator), and suicidal risk assessments (monitored bi-weekly). Any participant at immediate risk, will be referred to a higher level of care and discontinued from the study. A participant is also removed in case of an intercurrent illness, or because they require a new drug or therapeutic method that has demonstrated its efficacy in this indication (in this case, the withdrawal from the trial will occur as soon as the new therapeutic agent is introduced).

   Any study withdrawal is documented and specified until the trial exit. The investigators replace each early drop out (over enrollment). Missing data will be handled through maximum likelihood estimation in the primary analysis models, using predictors of missingness and drop-out. The investigators will conduct regular quality checks to maintain data quality throughout. In case of uninterpretable data, they will recruit a few additional participants to reach N=30 with analyzable neuroimaging and psychophysiological data. The investigators anticipate to recruit n=35 total participants to obtain N=30 participants with analyzable neuroimaging and psychophysiological data (anticipated dropout = 20%).
6. CONSIDERATIONS AND OBLIGATIONS:

   1. Standard Operating Procedures are created for all procedure which will address registry operations and analysis activities, such as patient recruitment, data collection, data management, data analysis, reporting for adverse events, and possible change management.
   2. Data are managed in a database administered by the sponsor, in accordance with the regulations in force. Data entry are performed by investigators at each center or any person on the task delegation list. A data dictionary is created that contains detailed descriptions of each variable used for data registry (e.g., information on variable source, normal (score) ranges). Data are identified only by participant codes, with all identifying information removed to protect confidentiality. Participant identity will not be revealed in any presentation or publication of results.
   3. In accordance with the French law, the participant may exercise their right to access and rectify data collected at any time. The participation of the person in the research as well as the modalities of the collection of his consent and the delivery of the information in order to collect it are specified in the participant's medical file. The sponsor will inform participants of the overall results of this research at the end of the study.
   4. Depending on level of risk and/or impact of the study defined by the sponsor, the data may be monitored randomly. In this case, a person mandated by the sponsor will monitor the data collected in the data collection booklet (verification from the patient's medical record). It is therefore the investigator's responsibility to give free access to all the medical records of the participants involved in the research (having signed a consent form).
   5. The investigator agrees to accept quality assurance audits by the sponsor or inspections by the health authorities.

ELIGIBILITY:
Inclusion Criteria:

* Must have lost a loved one (spouse, romantic partner, parent, child, sibling, close friend)
* Must have a score >29 on the Inventory of Complicated Grief (ICG)
* Clinical diagnosis of Prolonged Grief Disorder as assessed by the Structured Clinical Interview for Complicated Grief (SCI-CG)

Exclusion Criteria:

* History of a lifetime clinical diagnosis of schizophrenia
* History of a lifetime clinical diagnosis of bipolar disorder
* History of a lifetime clinical diagnosis of a psychotic disorder
* Current diagnosis of substance or alcohol use disorder within the past 12 months
* History of a neurologic disease, seizures, stroke or head injury resulting in prolonged loss of consciousness and/or neurological sequelae
* Current pregnancy as assessed by a urinary pregnancy test at screening during the Screening (week -4 until 0), Baseline (week 0) or Endpoint visit (week 8), or lack of use approved methods birth control for women of childbearing age
* Currently practice of mind-body techniques at least once a week (e.g., yoga) in the past 3 months
* Currently undergoing concomitant psychotherapy for grief (any psychotherapy)
* Left-handedness
* Current use of medications that would affect cerebral metabolism
* Any contraindications to Magnetic Resonance Imaging (MRI)
* Being under legal guardianship

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in Prolonged Grief Disorder (PGD) symptom severity from the pre-intervention baseline to the post-intervention endpoint visit. | Assessed during the pre-intervention baseline (week 0), post-intervention endpoint (week 8), and one-month follow-up visit (week 12).
  PGD symptom severity is assessed by the Inventory of Complicated Grief (ICG) questionnaire.

SECONDARY OUTCOMES:
Mean change in Prolonged Grief Disorder (PGD) symptom severity from the pre-intervention baseline to the post-intervention endpoint, and one-month follow-up visit. | Assessed during the pre-intervention baseline (week 0), post-intervention endpoint (week 8), and one-month follow-up visit (week 12).
  PGD symptom severity is assessed by the Structural Clinical Interview for Complicated Grief (SCI-CG).
Mean change in Posttraumatic Stress Disorder (PTSD) symptom severity in relation to the death, from the pre-intervention baseline to the post-intervention endpoint, and one-month follow-up visit. | Assessed during the pre-intervention baseline (week 0), post-intervention endpoint (week 8), and one-month follow-up visit (week 12).
  PTSD symptom severity is assessed by the PTSD Checklist for DSM-5 (PCL-5).
Mean change in Depression symptom severity from the pre-intervention baseline to the post-intervention endpoint, and one-month follow-up visit. | Assessed during the pre-intervention baseline (week 0), post-intervention endpoint (week 8), and one-month follow-up visit (week 12).
  Depression symptom severity is assessed by the Quick Inventory of Depressive Symptomatology (QIDS-SR).
Mean change in somatic complaints from the pre-intervention baseline to the post-intervention endpoint, and one-month follow-up visit. | Assessed during the pre-intervention baseline (week 0), post-intervention endpoint (week 8), and one-month follow-up visit (week 12).
  Somatic symptoms are assessed by the Medical Symptom Checklist (MSCL).
Mean change in the ability to cope with stress from the pre-intervention baseline to the post-intervention endpoint, and one-month follow-up visit. | Assessed during the pre-intervention baseline (week 0), post-intervention endpoint (week 8), and one-month follow-up visit (week 12).
  Coping ability with stress is assessed by the Measure of Current Status (MOCS).
Mean change in global symptom severity from the pre-intervention baseline to the post-intervention endpoint, and one-month follow-up visit. | Assessed during the pre-intervention baseline (week 0), post-intervention endpoint (week 8), and one-month follow-up visit (week 12).
  Global symptom severity is assessed by the Clinical Global Impressions of Severity scale (CGI-S).
Mean change in global symptom improvement from the mid-intervention midpoint to the post-intervention endpoint, and one-month follow-up visit. | Assessed during the mid-intervention midpoint (week 4), post-intervention endpoint (week 8), and one-month follow-up visit (week 12).
  Global symptom improvement is assessed by the Clinical Global Impressions of Improvement scale (CGI-I).
Mean change in skin conductance response rates to bereavement-related stress from the pre-intervention baseline to the post-intervention endpoint visit. | Assessed during the pre-intervention baseline (week 0) and post-intervention endpoint visit (week 8).
  Skin conductance response rates during the Script-Driven Imagery paradigm are measured as peripheral biomarkers of bereavement-related stress reactivity in the neuroimaging scanner.
Mean change in heart rate responses to bereavement-related stress from the pre-intervention baseline to the post-intervention endpoint visit. | Assessed during the pre-intervention baseline (week 0) and post-intervention endpoint visit (week 8).
  Heart rate responses during the Script-Driven Imagery paradigm are measured as peripheral biomarkers of bereavement-related stress reactivity in the neuroimaging scanner.
Mean change in skin conductance response rates during general stress from the pre-intervention baseline to the post-intervention endpoint visit. | Assessed during the pre-intervention baseline (week 0) and post-intervention endpoint visit (week 8).
  Skin conductance response rates during the Loud Tones paradigm are measured as peripheral biomarkers of general stress reactivity in the neuroimaging scanner.
Mean change in heart rate responses to general stress from the pre-intervention baseline to the post-intervention endpoint visit. | Assessed during the pre-intervention baseline (week 0) and post-intervention endpoint visit (week 8).
  Heart rate responses during the Loud Tones paradigm are measured as peripheral biomarkers of general stress reactivity in the neuroimaging scanner.
Mean change in Blood Oxygentation Level Dependent (BOLD brain activity) signals during bereavement-related stress from the pre-intervention baseline to the post-intervention endpoint visit. | Assessed during the pre-intervention baseline (week 0) and post-intervention endpoint visit (week 8).
  Blood Oxygentation Level Dependent (BOLD brain activity) signals during a Script-Driven Imagery paradigm are measured as neural biomarkers of bereavement-related stress reactivity in the neuroimaging scanner.
Mean change in brain Functional Connectivity during bereavement-related stress from the pre-intervention baseline to the post-intervention endpoint visit. | Assessed during the pre-intervention baseline (week 0) and post-intervention endpoint visit (week 8).
  Brain Functional Connectivity during a Script-Driven Imagery paradigm are measured as neural biomarkers of bereavement-related stress reactivity in the neuroimaging scanner.
Mean change in Blood Oxygentation Level Dependent (BOLD brain activity) signals during general stress from the pre-intervention baseline to the post-intervention endpoint visit. | Assessed during the pre-intervention baseline (week 0) and post-intervention endpoint visit (week 8).
  Blood Oxygentation Level Dependent (brain activity) signals during a Loud Tones paradigm are measured as neural biomarkers of general stress reactivity in the neuroimaging scanner.
Mean change in brain Functional Connectivity during general stress from the pre-intervention baseline to the post-intervention endpoint visit. | Assessed during the pre-intervention baseline (week 0) and post-intervention endpoint visit (week 8).
  Brain Functional Connectivity during a Loud Tones paradigm are measured as neural biomarkers of general stress reactivity in the neuroimaging scanner.

OTHER OUTCOMES:
Characteristics of the death. | Assessed during the screening visit (week-4 until 0).
  Charcteristics of the death are assessed as covariates and include the time since the loss, the type of death, the cause of death, and the relationship between the participant and the deceased.
The absence of diagnostic exclusion criteria and co-occurring Axis-I psychiatric disorders. | Assessed during the screening visit (week-4 until 0).
  Diagnoses is assessed by the Mini International Neuropsychiatric Interview (MINI).
Socio-demographic variables. | Assessed during the screening visit (week-4 until 0).
  Socio-demographic variables are assessed as potential Confounders for grief reactions and include age, sex, gender, socioeconomic status, educational level, racial and ethnic origins, menstrual cycle information, and handedness.
Self-reports of mood and bereavement-related stress responses. | Assessed during each imagery phase of the Script-Driven Imagery paradigm during the pre-intervention baseline (week 0) and post-intervention endpoint visit (week 8).
  Self-report mood and bereavement-related stress responses measured on 8-point Likert scales (range 0 "none" - 8 "a great deal") are assessed for vividness, valence related to control/dominance, happiness/pleasure, and excitement/ arousal of their imagery, as well as feelings of sadness, anger, fear, disgust, surprise, guilt, emotional pain and yearning for the deceased during each imagery phase of the Script-Driven Imagery paradigm in the neuroimaging scanner to check that the paradigm elicited the intended emotions.
Mean change in self-reports of mood and bereavement-related stress responses from the pre-intervention baseline to the post-intervention endpoint visit. | Assessed during each imagery phase of the Script-Driven Imagery paradigm, and from the pre-intervention baseline (week 0) to post-intervention endpoint visit (week 8).
  Self-report mood and bereavement-related stress responses measured on 8-point Likert scales (range 0 "none" - 8 "a great deal") are assessed for vividness, valence related to control/dominance, happiness/pleasure, and excitement/ arousal of their imagery, as well as feelings of sadness, anger, fear, disgust, surprise, guilt, emotional pain and yearning for the deceased during each imagery phase of the Script-Driven Imagery paradigm in the neuroimaging scanner.
Procedure-related time variables. | Assessed during the screening visit (week -4 until 0), baseline visit (week 0), midpoint visit (week 4), endpoint visit (week 8), follow-up visit (week 12), and 2-weekly safety checks (week 2, week 6).
  Procedure-related time variables are assessed as potential potential covariates and include time of arrival and end time during assessment visits.
Potential adverse events experienced by the participant. | Assessed during the screening visit (week -4 until 0), baseline visit (week 0), midpoint visit (week 4), endpoint visit (week 8), follow-up visit (week 12), and 2-weekly safety checks (week 2, week 6).
  Potential adverse events are assessed as safety check-in assessment using the Adverse Events Monitoring Form.
Suicidal risk experienced by the participant. | Assessed during the screening visit (week -4 until 0), baseline visit (week 0), midpoint visit (week 4), endpoint visit (week 8), follow-up visit (week 12), and 2-weekly safety checks (week 2, week 6).
  Suicidal risk is assessed as safety check-in assessment and will include the severity of a patient's suicidal ideation using the Clinician Suicide Assessment Checklist (CSAS).
Procedure-related comments | Assessed during the screening visit (week -4 until 0), baseline visit (week 0), midpoint visit (week 4), endpoint visit (week 8), follow-up visit (week 12), and 2-weekly safety checks (week 2, week 6).
  Procedure-related comments are assessed as any important notes or comments about the research procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Eric BUI, Professor, Principal Investigator — CHU de Caen, Université de Caen Normandie, INSERM U1237, PhIND; Annick Haelewyn-Razafimandimby, Associate Pr, Study Director — INSERM U1237, PhIND; Charlotte Hilberdink, Postdoc, Study Chair — INSERM U1237, PhIND
Locations (1):
- CHU de Caen et Université de Caen Normandie - Centre Esquirol Adult Psychiatry, Caen, Calvados, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benson H, Greenwood MM, Klemchuk H. The relaxation response: psychophysiologic aspects and clinical applications. Int J Psychiatry Med. 1975;6(1-2):87-98. doi: 10.2190/376W-E4MT-QM6Q-H0UM. PMID 773864
- [Background] Borysenko, J. (1988). Minding the Body Mending the Mind. New York, Bantam.
- [Background] Bowlby, J. (1980). Attachment and loss, volume 3: loss; sadness and depression.
- [Background] Bui E, Mauro C, Robinaugh DJ, Skritskaya NA, Wang Y, Gribbin C, Ghesquiere A, Horenstein A, Duan N, Reynolds C, Zisook S, Simon NM, Shear MK. THE STRUCTURED CLINICAL INTERVIEW FOR COMPLICATED GRIEF: RELIABILITY, VALIDITY, AND EXPLORATORY FACTOR ANALYSIS. Depress Anxiety. 2015 Jul;32(7):485-92. doi: 10.1002/da.22385. Epub 2015 Jun 9. PMID 26061724
- [Background] Bui E, Blackburn AM, Brenner LH, Laifer LM, Park ER, Fricchione GL, Sylvia LG. Military and Veteran Caregivers' Perspectives of Stressors and a Mind-Body Program. Issues Ment Health Nurs. 2018 Oct;39(10):850-857. doi: 10.1080/01612840.2018.1485796. Epub 2018 Sep 13. PMID 30212258
- [Background] Eric Bui, Ilana Ander & Clara Jaussaud. (2021). Grief in the time of COVID-19: An editorial, International Journal of Mental Health, 50:1, 1-3, DOI: 10.1080/00207411.2020.1870847
- [Background] Carson MA, Metzger LJ, Lasko NB, Paulus LA, Morse AE, Pitman RK, Orr SP. Physiologic reactivity to startling tones in female Vietnam nurse veterans with PTSD. J Trauma Stress. 2007 Oct;20(5):657-66. doi: 10.1002/jts.20218. PMID 17955532
- [Background] Currier JM, Neimeyer RA, Berman JS. The effectiveness of psychotherapeutic interventions for bereaved persons: a comprehensive quantitative review. Psychol Bull. 2008 Sep;134(5):648-661. doi: 10.1037/0033-2909.134.5.648. PMID 18729566
- [Background] Dawson, M.E., Schell, A.M., and Filion, D.L. (2017). The electrodermal system. In J.T. Cacioppo, L.G. Tassinary, G.G. Berntson (Eds.), Handbook of Psychophysiology, Cambridge University Press, New York, NY, pp. 217-243.
- [Background] Guy W. (1979). ECDEU Assessment Manual for Psychopharmacology. Rockville, MD, U.S. Department of Health, Education, and Welfare.
- [Background] Hoge EA, Bui E, Marques L, Metcalf CA, Morris LK, Robinaugh DJ, Worthington JJ, Pollack MH, Simon NM. Randomized controlled trial of mindfulness meditation for generalized anxiety disorder: effects on anxiety and stress reactivity. J Clin Psychiatry. 2013 Aug;74(8):786-92. doi: 10.4088/JCP.12m08083. PMID 23541163
- [Background] Hoge EA, Bui E, Palitz SA, Schwarz NR, Owens ME, Johnston JM, Pollack MH, Simon NM. The effect of mindfulness meditation training on biological acute stress responses in generalized anxiety disorder. Psychiatry Res. 2018 Apr;262:328-332. doi: 10.1016/j.psychres.2017.01.006. Epub 2017 Jan 26. PMID 28131433
- [Background] Hoge EA, Bui E, Mete M, Dutton MA, Baker AW, Simon NM. Mindfulness-Based Stress Reduction vs Escitalopram for the Treatment of Adults With Anxiety Disorders: A Randomized Clinical Trial. JAMA Psychiatry. 2023 Jan 1;80(1):13-21. doi: 10.1001/jamapsychiatry.2022.3679. PMID 36350591
- [Background] Kabat-Zinn, J. (1990). Full Catastrophe Living: Using the Wisdom of Your Body and Mind to Face Stress, Pain, and Illness, Bantam Dell.
- [Background] Kang, Y., Gruber, J., & Gray, J. R. (2013). Mindfulness and De-Automatization. Emotion Review, 5(2), 192-201. https://doi.org/10.1177/1754073912451629
- [Background] Khoury B, Lecomte T, Fortin G, Masse M, Therien P, Bouchard V, Chapleau MA, Paquin K, Hofmann SG. Mindfulness-based therapy: a comprehensive meta-analysis. Clin Psychol Rev. 2013 Aug;33(6):763-71. doi: 10.1016/j.cpr.2013.05.005. Epub 2013 Jun 7. PMID 23796855
- [Background] Lang PJ. Presidential address, 1978. A bio-informational theory of emotional imagery. Psychophysiology. 1979 Nov;16(6):495-512. doi: 10.1111/j.1469-8986.1979.tb01511.x. No abstract available. PMID 515293
- [Background] Latham AE, Prigerson HG. Suicidality and bereavement: complicated grief as psychiatric disorder presenting greatest risk for suicidality. Suicide Life Threat Behav. 2004 Winter;34(4):350-62. doi: 10.1521/suli.34.4.350.53737. PMID 15585457
- [Background] Laurie A, Neimeyer RA. African Americans in bereavement: grief as a function of ethnicity. Omega (Westport). 2008;57(2):173-93. doi: 10.2190/OM.57.2.d. PMID 18680889
- [Background] LeBlanc NJ, Unger LD, McNally RJ. Emotional and physiological reactivity in Complicated Grief. J Affect Disord. 2016 Apr;194:98-104. doi: 10.1016/j.jad.2016.01.024. Epub 2016 Jan 13. PMID 26803781
- [Background] Lichtenthal WG, Nilsson M, Kissane DW, Breitbart W, Kacel E, Jones EC, Prigerson HG. Underutilization of mental health services among bereaved caregivers with prolonged grief disorder. Psychiatr Serv. 2011 Oct;62(10):1225-9. doi: 10.1176/ps.62.10.pss6210_1225. PMID 21969652
- [Background] Marchand WR. Neural mechanisms of mindfulness and meditation: Evidence from neuroimaging studies. World J Radiol. 2014 Jul 28;6(7):471-9. doi: 10.4329/wjr.v6.i7.471. PMID 25071887
- [Background] Moon JR, Kondo N, Glymour MM, Subramanian SV. Widowhood and mortality: a meta-analysis. PLoS One. 2011;6(8):e23465. doi: 10.1371/journal.pone.0023465. Epub 2011 Aug 17. PMID 21858130
- [Background] Newson RS, Boelen PA, Hek K, Hofman A, Tiemeier H. The prevalence and characteristics of complicated grief in older adults. J Affect Disord. 2011 Jul;132(1-2):231-8. doi: 10.1016/j.jad.2011.02.021. Epub 2011 Mar 12. PMID 21397336
- [Background] O'Connor MF. Immunological and neuroimaging biomarkers of complicated grief. Dialogues Clin Neurosci. 2012 Jun;14(2):141-8. doi: 10.31887/DCNS.2012.14.2/mfoconnor. PMID 22754286
- [Background] O'Connor MF, Wellisch DK, Stanton AL, Eisenberger NI, Irwin MR, Lieberman MD. Craving love? Enduring grief activates brain's reward center. Neuroimage. 2008 Aug 15;42(2):969-72. doi: 10.1016/j.neuroimage.2008.04.256. Epub 2008 May 10. PMID 18559294
- [Background] Oltjenbruns KA. Ethnicity and the grief response: Mexican American versus Anglo American college students. Death Stud. 1998;22(2):141-55. doi: 10.1080/074811898201641. PMID 10182423
- [Background] Orr SP, Pitman RK, Lasko NB, Herz LR. Psychophysiological assessment of posttraumatic stress disorder imagery in World War II and Korean combat veterans. J Abnorm Psychol. 1993 Feb;102(1):152-9. doi: 10.1037//0021-843x.102.1.152. PMID 8436691
- [Background] Park ER, Traeger L, Vranceanu AM, Scult M, Lerner JA, Benson H, Denninger J, Fricchione GL. The development of a patient-centered program based on the relaxation response: the Relaxation Response Resiliency Program (3RP). Psychosomatics. 2013 Mar-Apr;54(2):165-74. doi: 10.1016/j.psym.2012.09.001. Epub 2013 Jan 22. PMID 23352048
- [Background] Pole N, Neylan TC, Best SR, Orr SP, Marmar CR. Fear-potentiated startle and posttraumatic stress symptoms in urban police officers. J Trauma Stress. 2003 Oct;16(5):471-9. doi: 10.1023/A:1025758411370. PMID 14584631
- [Background] Prigerson HG, Maciejewski PK, Reynolds CF 3rd, Bierhals AJ, Newsom JT, Fasiczka A, Frank E, Doman J, Miller M. Inventory of Complicated Grief: a scale to measure maladaptive symptoms of loss. Psychiatry Res. 1995 Nov 29;59(1-2):65-79. doi: 10.1016/0165-1781(95)02757-2. PMID 8771222
- [Background] Prigerson HG, Bierhals AJ, Kasl SV, Reynolds CF 3rd, Shear MK, Day N, Beery LC, Newsom JT, Jacobs S. Traumatic grief as a risk factor for mental and physical morbidity. Am J Psychiatry. 1997 May;154(5):616-23. doi: 10.1176/ajp.154.5.616. PMID 9137115
- [Background] Rauch SAM, Kim HM, Lederman S, Sullivan G, Acierno R, Tuerk PW, Simon NM, Venners MR, Norman SB, Allard CB, Porter KE, Martis B, Bui E, Baker AW; PROGrESS Team. Predictors of Response to Prolonged Exposure, Sertraline, and Their Combination for the Treatment of Military PTSD. J Clin Psychiatry. 2021 Jun 15;82(4):20m13752. doi: 10.4088/JCP.20m13752. PMID 34133087
- [Background] Reynolds CF 3rd, Miller MD, Pasternak RE, Frank E, Perel JM, Cornes C, Houck PR, Mazumdar S, Dew MA, Kupfer DJ. Treatment of bereavement-related major depressive episodes in later life: a controlled study of acute and continuation treatment with nortriptyline and interpersonal psychotherapy. Am J Psychiatry. 1999 Feb;156(2):202-8. doi: 10.1176/ajp.156.2.202. PMID 9989555
- [Background] Rostila M, Saarela J, Kawachi I, Hjern A. Testing the anniversary reaction: causal effects of bereavement in a nationwide follow-up study from Sweden. Eur J Epidemiol. 2015 Mar;30(3):239-47. doi: 10.1007/s10654-015-9989-5. Epub 2015 Jan 17. PMID 25595319
- [Background] Rush AJ, Trivedi MH, Ibrahim HM, Carmody TJ, Arnow B, Klein DN, Markowitz JC, Ninan PT, Kornstein S, Manber R, Thase ME, Kocsis JH, Keller MB. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry. 2003 Sep 1;54(5):573-83. doi: 10.1016/s0006-3223(02)01866-8. PMID 12946886
- [Background] Samuelson M, Foret M, Baim M, Lerner J, Fricchione G, Benson H, Dusek J, Yeung A. Exploring the effectiveness of a comprehensive mind-body intervention for medical symptom relief. J Altern Complement Med. 2010 Feb;16(2):187-92. doi: 10.1089/acm.2009.0142. PMID 20180692
- [Background] Sbarra DA, Hazan C. Coregulation, dysregulation, self-regulation: an integrative analysis and empirical agenda for understanding adult attachment, separation, loss, and recovery. Pers Soc Psychol Rev. 2008 May;12(2):141-67. doi: 10.1177/1088868308315702. PMID 18453476
- [Background] Selye, H. (1956). The stress of life. McGraw-Hill.
- [Background] Shear K, Frank E, Houck PR, Reynolds CF 3rd. Treatment of complicated grief: a randomized controlled trial. JAMA. 2005 Jun 1;293(21):2601-8. doi: 10.1001/jama.293.21.2601. PMID 15928281
- [Background] Shear MK, Ghesquiere A, Glickman K. Bereavement and complicated grief. Curr Psychiatry Rep. 2013 Nov;15(11):406. doi: 10.1007/s11920-013-0406-z. PMID 24068457
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Shin LM, Orr SP, Carson MA, Rauch SL, Macklin ML, Lasko NB, Peters PM, Metzger LJ, Dougherty DD, Cannistraro PA, Alpert NM, Fischman AJ, Pitman RK. Regional cerebral blood flow in the amygdala and medial prefrontal cortex during traumatic imagery in male and female Vietnam veterans with PTSD. Arch Gen Psychiatry. 2004 Feb;61(2):168-76. doi: 10.1001/archpsyc.61.2.168. PMID 14757593
- [Background] Shor E, Roelfs DJ, Curreli M, Clemow L, Burg MM, Schwartz JE. Widowhood and mortality: a meta-analysis and meta-regression. Demography. 2012 May;49(2):575-606. doi: 10.1007/s13524-012-0096-x. PMID 22427278
- [Background] Simon NM, Hofmann SG, Rosenfield D, Hoeppner SS, Hoge EA, Bui E, Khalsa SBS. Efficacy of Yoga vs Cognitive Behavioral Therapy vs Stress Education for the Treatment of Generalized Anxiety Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2021 Jan 1;78(1):13-20. doi: 10.1001/jamapsychiatry.2020.2496. PMID 32805013
- [Background] Thompson LW, Breckenridge JN, Gallagher D, Peterson J. Effects of bereavement on self-perceptions of physical health in elderly widows and widowers. J Gerontol. 1984 May;39(3):309-14. doi: 10.1093/geronj/39.3.309. PMID 6715808
- [Background] Vranceanu AM, Riklin E, Merker VL, Macklin EA, Park ER, Plotkin SR. Mind-body therapy via videoconferencing in patients with neurofibromatosis: An RCT. Neurology. 2016 Aug 23;87(8):806-14. doi: 10.1212/WNL.0000000000003005. Epub 2016 Jul 22. PMID 27449066
- [Background] Waller A, Turon H, Mansfield E, Clark K, Hobden B, Sanson-Fisher R. Assisting the bereaved: A systematic review of the evidence for grief counselling. Palliat Med. 2016 Feb;30(2):132-48. doi: 10.1177/0269216315588728. Epub 2015 Sep 28. PMID 26415735
- [Background] Wittouck C, Van Autreve S, De Jaegere E, Portzky G, van Heeringen K. The prevention and treatment of complicated grief: a meta-analysis. Clin Psychol Rev. 2011 Feb;31(1):69-78. doi: 10.1016/j.cpr.2010.09.005. Epub 2010 Sep 24. PMID 21130937
- [Background] Zisook S, Shear K. Grief and bereavement: what psychiatrists need to know. World Psychiatry. 2009 Jun;8(2):67-74. doi: 10.1002/j.2051-5545.2009.tb00217.x. PMID 19516922
- [Background] American Psychiatric Association, DSM-5 Task Force. (2013). Diagnostic and statistical manual of mental disorders: DSM-5™ (5th ed.). American Psychiatric Publishing, Inc.. https://doi.org/10.1176/appi.books.9780890425596
- See also: Weathers, F., B. Litz, T. Keane, P. Palmieri, B. Marx and P. Schnurr (2013). The PTSD Checklist for DSM-5 (PCL-5). Scale available from the National Center for PTSD. — https://www.ptsd.va.gov/professional/assessment/adult-sr/ptsd-checklist.asp